CLINICAL TRIAL: NCT02407795
Title: A RAndomized Trial Comparing COnventional With STereotactic Radiotherapy for Pain Reduction and Quality of Life in Spinal Metastases (RACOST-trial)
Brief Title: Conventional With Stereotactic Radiotherapy for Pain Reduction and Quality of Life in Spinal Metastases
Acronym: RACOST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: very slow inclusion
Sponsor: Radboud University Medical Center (Other)
Collaborators: Koningin Wilhelmina Fonds (Other); Maastro Clinic, The Netherlands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NL45994.091.14
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Spinal Metastases
Keywords: stereotactic radiotherapy; pain reduction; quality of life
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): Conventional radiotherapy, 1x8Gy
  Interventions: Radiation: conventional radiotherapy
- Arm 2 (Experimental): Stereotactic radiotherapy, 1x20Gy
  Interventions: Radiation: stereotactic radiotherapy

INTERVENTIONS:
Radiation: conventional radiotherapy — 1x8Gy
  Arms: Arm 1
Radiation: stereotactic radiotherapy — 1x20Gy or equivalent dose fractionation schedule
  Arms: Arm 2

SUMMARY:
A randomized, multicentre, phase III study comparing conventional radiotherapy (1x8Gy) with stereotactic radiotherapy (1x20Gy) for pain reduction and quality of life in spinal metastases.

DETAILED DESCRIPTION:
Study population: patients with painful spinal metastases from solid tumors without spinal cord compression or cord instability.

Objective: This study will test the hypothesis that stereotactic radiotherapy gives a better and longer lasting reduction of pain, local control and therewith a better quality of life. This in order to optimize and to individualize the treatment options for the patient.

Study design: Complaints due to pain will be analysed using the validated Dutch Brief Pain Inventory (BPI) and side-effects will be recorded using the Common Toxicity Criteria for Adverse Events (CTCAE). In addition to this the quality of life will be analysed using the EORTC QOL-C15-PAL and EORTC QLQ-BM22 questionnaires. For analysis of cost-effectiveness the EQ-5D will be used.

ELIGIBILITY:
Inclusion Criteria:

* solid tumor with radiological diagnosis of spinal metastases
* pain score minimum 2 on 11-point scale
* maximum of 2 consecutive or noncontiguous spinal vertebra involved by tumor at current level of interest
* No or mild neurological signs (radiculopathy, dermatomal sensory change and muscle strength of involved extremity)
* Karnofsky performance ≥60
* WHO ≤2
* life expectancy > 6 weeks
* age ≥18
* non-pregnant, non-lactating female patients

Exclusion Criteria:

* history of previous radiotherapy to the spine at current level of interest
* spinal instability or neurological deficit
* pathological fracture or impending fracture needing fixation
* prior surgery to the spine at current level of interest
* clinical signs of spinal cord compression or severe neurological deficits
* patients with a pacemaker such that MRI cannot be performed or the treatment cannot be delivered safely
* patients unable to undergo MRI
* earlier nuclear medicine treatment
* pregnancy
* altered mental status that would prohibit the understanding and giving of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Pain reduction measured by the Dutch Brief Pain Inventory (BPI) questionnaire | At six weeks since baseline
  Pain is self-reported and measured by the validated Dutch Brief Pain Inventory (BPI) questionnaire

SECONDARY OUTCOMES:
Comparison of time to pain response | pain response is calculated from the date of randomization at day 0-14, week 4, 6, and month 2, 3, 4, 6, 9, and 12
  Pain is self-reported and measured by the validated Dutch Brief Pain Inventory (BPI) questionnaire
Duration of pain relief | Pain relief is calculated from the date of randomization at day 0-14, week 4, 6, and month 2, 3, 4, 6, 9, and 12
  Pain is self-reported and measured by the validated Dutch Brief Pain Inventory (BPI) questionnaire
Quality of life | Quality of life is calculated from the date of randomization at day 0, 7, 14, week 4, 6, and month 2, 3, 4, 6, 9, and 12
  EORTC QOL-C15-PAL and EORTC QLQ-BM22 questionnaires
Toxicity measured by CTCAE 4.0 questionnaire | up to months 12
  Toxicity measuredCTCAE 4.0 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: P Braam, MD, Principal Investigator — Radboudumc Nijmegen
Locations (6):
- Netherlands (6):
  - Radiotherapiegroep Arnhem, Arnhem
  - Radiotherapiegroep Deventer, Deventer
  - MAASTRO clinic, Maastricht
  - Radboudumc Nijmegen, Nijmegen
  - Medisch Centrum Haaglanden, The Hague
  - Isala, Zwolle

REFERENCES:
- [Derived] Braam P, Lambin P, Bussink J. Stereotactic versus conventional radiotherapy for pain reduction and quality of life in spinal metastases: study protocol for a randomized controlled trial. Trials. 2016 Feb 2;17:61. doi: 10.1186/s13063-016-1178-7. PMID 26829933